CLINICAL TRIAL: NCT00306072
Title: Effect of Different Doses of Salacinol Extract on Glycemic and Insulinemic Response in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ross Products (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CP-SRDB28
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2006-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Drug: nutritional herbal extract from Salacia oblonga

SUMMARY:
The purpose of this study is to evaluate two levels of the herbal extract Salacia oblonga (salacinol) on postprandial glycemia and insulinemia in patients with Type 2 diabetes after ingestion of a high-carbohydrate control meal.

DETAILED DESCRIPTION:
Although we have generated a good quantity of animal and human data on the salacinol extract, we have not explored the effect of the salacinol extract on postprandial glycemia or insulinemia in patients with type 2 diabetes.

We planned to study 66 patients with diabetes in this multicenter, randomized, double-blind, three-treatment, crossover study. While in a fasted state, subjects were to consume one of the following three meals: a standard liquid meal containing 110 g carbohydrate, 18 g protein, 12 g fat, and 620 kilocalories (Control); Control plus 240 mg Salacia oblonga extract; and Control plus 480 mg Salacia oblonga extract. Postprandial serum glucose and serum insulin samples were to be analyzed for 180 min.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has type 2 diabetes mellitus verified by prescription of oral antihyperglycemic medications.
2. Subject is 18 to 75 years of age, inclusively.
3. Subject is male or a nonpregnant, nonlactating female, at least six weeks postpartum. A urine pregnancy test is required for all female subjects unless subject has had a hysterectomy, tubal ligation, or is > 2 years postmenopausal.
4. Subject has a body mass index (BMI) of 18 - 35 kg/m2.
5. Subject has voluntarily signed and dated an informed consent form, approved by an Independent Ethics Committee/Institutional Review Board and provided HIPAA (or other applicable privacy regulation) authorization prior to any participation in the study.

Exclusion Criteria:

1. Subject uses exogenous insulin for glucose control.
2. Subject states that he/she has an infection (requiring medication or hospitalization).
3. Subject states that he/she has current hepatic disease.
4. Subject states that he/she has had surgery, or corticosteroid treatment in the last 3 months or antibiotics in the last 3 weeks.
5. Subject has a first-degree relative enrolled in the current study.
6. Subject states that he/she has an active malignancy (subjects with cutaneous malignancies, other than melanoma, may be included in the study).
7. Subject states that he/she has had a significant cardiovascular event < 12 weeks prior to study entry.
8. Subject states that he/she has end stage organ failure, including clinically advanced renal disease as assessed by the study physician.
9. Subject states that he/she is status post-organ transplantation.
10. Subject states that he/she has a chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV.
11. Subject states that he/she has active metabolic or gastrointestinal diseases that may interfere with nutrient absorption, metabolism, or excretion, excluding diabetes.
12. As determined by the study physician, subject is taking daily medications or dietary supplements at doses that would interfere with nutrient absorption, metabolism, excretion or gastric motility.
13. Subject states that he/she has an allergy or intolerance to any ingredient found in the study products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82
Dates: Start 2005-06; Study Completion 2005-09

PRIMARY OUTCOMES:
The primary variable to be measured was positive AUC (0-180 minutes) for plasma glucose.

SECONDARY OUTCOMES:
The secondary variables to be measured were:
· Positive AUC (0 to 120 minutes) for plasma and serum glucose and positive AUC (0 to 180 minutes) for serum glucose
· Adjusted peak value for plasma and serum glucose
· Adjusted peak value for serum insulin
· Positive AUC 0-180 (0 to 120) minutes for serum insulin

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Williams, MPH, Study Director — Ross Products Division of Abbott Laboratories
Locations (2):
- United States (2):
  - Radiant Research, Edina, Minnesota
  - Radiant Research, Cincinnati, Ohio

REFERENCES:
- [Background] Hogan P, Dall T, Nikolov P; American Diabetes Association. Economic costs of diabetes in the US in 2002. Diabetes Care. 2003 Mar;26(3):917-32. doi: 10.2337/diacare.26.3.917. PMID 12610059
- [Background] Collene AL, Hertzler SR, Williams JA, Wolf BW. Effects of a nutritional supplement containing Salacia oblonga extract and insulinogenic amino acids on postprandial glycemia, insulinemia, and breath hydrogen responses in healthy adults. Nutrition. 2005 Jul-Aug;21(7-8):848-54. doi: 10.1016/j.nut.2004.11.018. PMID 15975493
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Ghavami A, Johnston BD, Pinto BM. A new class of glycosidase inhibitor: synthesis of salacinol and its stereoisomers. J Org Chem. 2001 Apr 6;66(7):2312-7. doi: 10.1021/jo001444g. PMID 11281771
- [Background] Heacock PM, Hertzler SR, Williams JA, Wolf BW. Effects of a medical food containing an herbal alpha-glucosidase inhibitor on postprandial glycemia and insulinemia in healthy adults. J Am Diet Assoc. 2005 Jan;105(1):65-71. doi: 10.1016/j.jada.2004.11.001. PMID 15635348
- [Background] Matsuda H, Murakami T, Yashiro K, Yamahara J, Yoshikawa M. Antidiabetic principles of natural medicines. IV. Aldose reductase and qlpha-glucosidase inhibitors from the roots of Salacia oblonga Wall. (Celastraceae): structure of a new friedelane-type triterpene, kotalagenin 16-acetate. Chem Pharm Bull (Tokyo). 1999 Dec;47(12):1725-9. doi: 10.1248/cpb.47.1725. PMID 10748716
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Wolf BW, Weisbrode SE. Safety evaluation of an extract from Salacia oblonga. Food Chem Toxicol. 2003 Jun;41(6):867-74. doi: 10.1016/s0278-6915(03)00038-3. PMID 12738192
- [Background] Wolever TM, Jenkins DJ, Jenkins AL, Josse RG. The glycemic index: methodology and clinical implications. Am J Clin Nutr. 1991 Nov;54(5):846-54. doi: 10.1093/ajcn/54.5.846. PMID 1951155
- See also: Information in the diabetes fact sheet was valuable to the process of writing the study protocol. The fact sheet contains current prevalence data for diabetes in the US. — http://www.diabetes.org/diabetes-basics/diabetes-statistics/